CLINICAL TRIAL: NCT05739071
Title: JING SI HERBAL TEA in the Treatment of Lower Urinary Tract Symptoms After Intravesical Therapy in Patients With Bladder Cancer
Brief Title: JING SI HERBAL TEA and Urinary Tract Symptoms in Bladder Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-XD-132
Record Dates: First submitted 2023-01-13; First posted 2023-02-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lower Urinary Tract Symptoms; Intravenous Drug Usage; Bladder Cancer; Herbal Interaction
Keywords: Intravesical installaion; Bladder cancer; Lower urinary tract symptoms; JING SI HERBAL TEA
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Double Blind (patients and attending physicians), parallel design Experimental group: JING SI HERBAL TEA, twice a day, every time 1 sachet for 3 days after each intravesical installation Control group: Placebo, twice a day, every time 1 sachet for 3 days after each intravesical installation
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomly assigned into the two groups with equal number. The JING SI HERBAL TEA and placebo have the same outer packaging. One dedicated researcher will be responsible for random allocation and administration, neither the patients nor the attending physicians (responsible for recording symptoms) knows the correct grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (group 1) (Experimental): This group will receive two sachets of JING SI HERBAL TEA a day (one in the morning and one in the evening).
  Interventions: Dietary Supplement: JING SI HERBAL TEA
- Control (group 2) (Placebo Comparator): This group will receive two sachets of placebo a day (same way as group 1).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: JING SI HERBAL TEA — JING SI HERBAL TEA is a food, contain with herbal extracts
  Arms: Experimental (group 1)
Dietary Supplement: Placebo — Placebo will have the same appearance as JING SI HERBAL TEA
  Arms: Control (group 2)

SUMMARY:
To identify the effects of JING SI HERBAL TEA in the treatment of lower urinary tract symptoms after intravesical therapy in patients with bladder cancer.

DETAILED DESCRIPTION:
The patients with bladder cancer usually required trans urethral resection of bladder tumor (TUR-BT). Post-operative intravesical installation therapy is standard therapy. However, new onset lower urinary tract symptoms often occurred after these installation therapies. JING SI HERBAL TEA is a food contain of many herbal extracts with anti-inflammation effects. The current study is to find out the effects of JING SI HERBAL TEA in the treatment of this condition.

The patients will be divided into two groups by randomly assigned (estimated case number=100, experimental: control = 1: 1). The first group will receive two sachets of JING SI HERBAL TEA a day (one in the morning and one in the evening). The second group will receive two sachets of placebo a day (same way as group 1). The therapy will be three days after each intravesical installation therapies.

The outcome evaluations will use the American Urological Association Symptom Index and 12-Item Short Form Survey (SF-12). The baseline symptoms will be recorded before the first intravesical therapy. Patients will be asked to fill out the questionnaire every week (the same time for the next installation). Every other standard cancer therapies will not be will not be affected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis bladder cancer
* Under intravesical installation therapy

Exclusion Criteria:

* Patients under 20 years old or greater than 100 years old
* Women with pregnancy or breastfeeding plans
* Bladder cancer are being treated in another hospital
* Had admitted due to other disease in the past 3 months
* Unable to understand the questionnaire

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms | The outcome evaluation will be at the following time points: 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks and 6 weeks
  Change from baseline score at the following time will be recorded. The American urological association symptom index is a 7-item self report measure to assess the urinary symptoms. The score range from 0 to 35, the higher the severity.

SECONDARY OUTCOMES:
Life quality | The outcome evaluation will be at the following time points: 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks and 6 weeks
  Change from baseline score at the following time will be recorded. The 12-item shor form survey is a general health questionaire for life quality evaluation. The higher the value obtained, the more significant the impact on life.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Wu, bachelor, Study Director — Taichung Tzu Chi Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Taipei branch, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The JING SI HERBAL TEA and Placebo are provided by the Tzu Chi Medical Foundation. We can not determining whether there are sufficient materials to provide the other participants